CLINICAL TRIAL: NCT01203319
Title: The Immunogenicity and Safety of 60mcg and 30mcg Recombinant Hepatitis B Vaccines in People Aged 16 and Older Who Failed to Respond to Routine Administration of 10mcg Recombinant Hepatitis B Vaccines
Brief Title: The Immunogenicity and Safety of 60mcg/30mcg Recombinant Hepatitis B Vaccines in People Who Failed to Respond to Routine Administration of Hepatitis B Vaccines
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Shenzhen Kangtai Biological Products Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KT0003
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Results first posted 2012-04-23 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Hepatitis b
Keywords: immunogenicity; safety; recombinant hepatitis B vaccine; nonresponders
MeSH Terms: conditions — Hepatitis B | interventions — Hepatitis B Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 60mcg/1.0ml recombinant hepatitis B vaccine (Experimental): 600 participants aged 16 and older who failed to respond to routine administration of 10mcg recombinant hepatitis B vaccines to receive 60mcg/1.0ml recombinant hepatitis B vaccines on day 0, 30 and 60.
  Interventions: Biological: 60mcg/1.0ml recombinant hepatitis B vaccine
- 30mcg/1.0ml recombinant hepatitis B vaccine (Experimental): 600 participants aged 16 and older who failed to respond to routine administration of 10mcg recombinant hepatitis B vaccines to receive 30mcg/1.0ml recombinant hepatitis B vaccines on day 0, 30 and 60.
  Interventions: Biological: 30mcg/1.0ml recombinant hepatitis B vaccine
- 10mcg/1.0ml recombinant hepatitis B vaccine (Placebo Comparator): 300 participants aged 16 and older who failed to respond to routine administration of 10mcg recombinant hepatitis B vaccines to receive 10mcg/1.0ml recombinant hepatitis B vaccines on day 0, 30 and 60.
  Interventions: Biological: 10mcg/1.0ml recombinant hepatitis B vaccine

INTERVENTIONS:
Biological: 60mcg/1.0ml recombinant hepatitis B vaccine — to receive 60mcg/1.0ml recombinant HBV vaccines on day 0, 30 and 60
  Arms: 60mcg/1.0ml recombinant hepatitis B vaccine
Biological: 30mcg/1.0ml recombinant hepatitis B vaccine — to receive 30mcg/1.0ml recombinant hepatitis B vaccines on day 0, 30 and 60.
  Arms: 30mcg/1.0ml recombinant hepatitis B vaccine
Biological: 10mcg/1.0ml recombinant hepatitis B vaccine — to receive 10mcg/1.0ml recombinant hepatitis B vaccines on day 0, 30 and 60
  Arms: 10mcg/1.0ml recombinant hepatitis B vaccine

SUMMARY:
This study is an expanded Phase 2/Phase 3 clinical trial base on the safety data obtained from the phase 1 clinical trial. The purpose of this study is to further evaluate the immunogenicity and safety of 60mcg/30mcg recombinant hepatitis B vaccines in people aged 16 and older who failed to respond to routine administration of 10mcg recombinant hepatitis B vaccines and to explore the optimizing immunizing dose and immune procedure.

DETAILED DESCRIPTION:
The most effective method to prevent hepatitis B virus infection is to receive the vaccination of hepatitis b vaccine to get the protective antibody anti-HBs. Both the blood-derived hepatitis B vaccine and the recombinant hepatitis B vaccines have been proved to be effective and safe since the application in 1981 and 1989 respectively. Previous passive or active immunization testes indicated that the lowest effective level of anti-HBs for prevention of infection is 10mIU/ml. However there are still some recipients can't generate expected level of anti-HBs after the vaccinations. In adults, there are 5% to 10% recipients will failed to respond to routine administration of 10mcg recombinant hepatitis B vaccines, and those nonresponders are susceptible population even after the vaccinations. In this study, a recipient whose peak period (1 month after vaccination) levels of anti-HBs is lower than 10mIU/ml after finishing the vaccinations of 3 dose 10mcg hepatitis b vaccines is called nonresponders.

Nowadays, a lot tests are conducted on nonresponders to help them generate the protective antibody anti-HBs, including increase the antigen dosage of vaccines, increase the injections of vaccines, change the route of inoculation and the use of adjuvant. Unfortunately, these previous studies can not get coincident and persuasive outcomes due to the small sample size and poor representativeness. This study is plan to evaluate the immunogenicity and safety of 60mcg/30mcg recombinant hepatitis B vaccines in people aged 16 and older who failed to respond to routine administration of 10mcg recombinant hepatitis B vaccines and to provide the scientific evidences for the revaccination strategy in China.

ELIGIBILITY:
Inclusion Criteria :

Filter period: The subjects to receive first 10mcg recombinant hepatitis B vaccines:

* Healthy subjects aged 16 and older as established by medical history and clinical examination
* The subjects or their guardians are able to understand and sign the informed consent
* Had never received the hepatitis B vaccines
* Subjects who can and will comply with the requirements of the protocol

Revaccination period: The nonresponders to receive first 60mcg recombinant hepatitis B vaccines:

* Healthy subjects aged 16 and older as established by medical history and clinical examination
* The subjects or their guardians are able to understand and sign the informed consent
* After the routine administration of 10mcg hepatitis B vaccines, the peak period levels of anti-HBs is lower than 10mIU/ml
* Subjects with temperature <37.1°C on axillary setting
* Subjects who can and will comply with the requirements of the protocol

Exclusion Criteria:

Filter period: The subjects to receive first 10mcg recombinant hepatitis B vaccines:

* Subject that has a medical history of any of the following: allergic history, or allergic to any ingredient of vaccine
* Family history of seizures or progressive neurological disease
* Family history of congenital or hereditary immunodeficiency
* Women of pregnancy, lactation or about to be pregnant in 60 days
* Autoimmune disease or immunodeficiency
* Bleeding disorder diagnosed by a doctor or significant bruising or bleeding difficulties with IM injections or blood draws
* Any prior administration of administration of immunoglobulins

Filter period: The subjects to receive second or/and third 10mcg recombinant hepatitis B vaccines:

* Any reaction or hypersensitivity to the recombinant hepatitis B vaccines after the vaccinations
* Serious adverse reactions to vaccines
* Active infections
* Subjects who want to quit the study
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives

Revaccination period: The nonresponders to receive first 60mcg recombinant hepatitis B vaccines:

* Qualitative test of Anti-HBs, HBsAg or Anti-HBc on serum is positive
* Any reaction or hypersensitivity to the recombinant hepatitis B vaccines after the vaccinations
* Family history of seizures or progressive neurological disease
* Family history of congenital or hereditary immunodeficiency
* Women of pregnancy, lactation or about to be pregnant in 60 days
* Autoimmune disease or immunodeficiency
* Bleeding disorder diagnosed by a doctor or significant bruising or bleeding difficulties with IM injections or blood draws
* Any prior administration of immunoglobulins, any other vaccines or experimental drugs in the last 7days
* Any active infections and received any antibiotic or anti-virus treatments in the last 7 days
* Had a fever in the last 3 days, with temperature ≥37.1°C
* Participate in another clinical trials
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives

Revaccination period: The nonresponders to receive second or/and third 60mcg recombinant hepatitis B vaccines:

* Any reaction or hypersensitivity to the recombinant hepatitis B vaccines after the vaccinations
* Serious adverse reactions to vaccines
* Active infections
* Subjects who want to quit the study
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1091 (Actual)
Dates: Start 2006-11; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Cai Zhu, Master, Principal Investigator — Jiangsu Provincial Center for Diseases Control and Prevention

REFERENCES:
- [Derived] Pan HX, Zeng Y, Song XF, Zhang YJ, Xu K, Liang ZL, Zhu FC. Immune response to hepatitis B vaccine with high antigen content in non-responders after standard primary vaccination in Chinese adults. Vaccine. 2014 Jun 17;32(29):3706-12. doi: 10.1016/j.vaccine.2014.02.094. Epub 2014 Mar 27. PMID 24681228

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 60mcg/1.0ml Recombinant Hepatitis B Vaccine | 30mcg/1.0ml Recombinant Hepatitis B Vaccine | 10mcg/1.0ml Recombinant Hepatitis B Vaccine
Started | 434 | 435 | 222
Completed | 428 | 426 | 217
Not Completed | 6 | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 60mcg/1.0ml Recombinant Hepatitis B Vaccine | 30mcg/1.0ml Recombinant Hepatitis B Vaccine | 10mcg/1.0ml Recombinant Hepatitis B Vaccine | Total
Number analyzed (Participants) | 434 | 435 | 222 | 1091
Age Continuous [Mean (Full Range); unit: years] | 42.7 [16 to 60] | 43.3 [16 to 60] | 42.6 [16 to 60] | 43.0 [16 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 226 | 220 | 115 | 561
  Male | 208 | 215 | 107 | 530

OUTCOME MEASURES:

1. Primary Outcome: Immunogenicity of Recombinant Hepatitis B Vaccines in Nonresponders
Description: Quantitative detection of anti-HBs using ratio-immunity method on serum obtained one month after second vaccination
Time Frame: one month after the second vaccination
Population: Accroding to Protocol set
Measure: Number; unit: participants
Arm/Group | 60mcg/1.0ml Recombinant Hepatitis B Vaccine | 30mcg/1.0ml Recombinant Hepatitis B Vaccine | 10mcg/1.0ml Recombinant Hepatitis B Vaccine
Number analyzed (Participants) | 428 | 426 | 217
participants | 394 [93.7 to 97.7] | 371 [89.6 to 94.8] | 180

2. Primary Outcome: Immunogenicity of Recombinant Hepatitis B Vaccines in Nonresponders
Description: Quantitative detection of anti-HBs using ratio-immunity method on serum obtained one month after third vaccination
Time Frame: one month after the third vaccination
Measure: Number; unit: participants
Arm/Group | 60mcg/1.0ml Recombinant Hepatitis B Vaccine | 30mcg/1.0ml Recombinant Hepatitis B Vaccine | 10mcg/1.0ml Recombinant Hepatitis B Vaccine
Number analyzed (Participants) | 428 | 426 | 217
participants | 411 | 394 | 187

3. Secondary Outcome: Immunogenicity of Recombinant Hepatitis B Vaccines in Nonresponders
Description: Quantitative detection of anti-HBs using ratio-immunity method on serum obtained one month after first vaccination
Time Frame: one month after the first vaccination
Measure: Number; unit: participants
Arm/Group | 60mcg/1.0ml Recombinant Hepatitis B Vaccine | 30mcg/1.0ml Recombinant Hepatitis B Vaccine | 10mcg/1.0ml Recombinant Hepatitis B Vaccine
Number analyzed (Participants) | 428 | 426 | 217
participants | 367 | 331 | 158

4. Secondary Outcome: the Safety of Recombinant Hepatitis B Vaccines in Nonresponders
Description: assessment of the local and systemic adverse reaction within the first 30 days after first vaccination
Time Frame: within the first 30 days after first vaccination
Reporting Status: Not Posted

5. Secondary Outcome: the Safety of Recombinant Hepatitis B Vaccines in Nonresponders
Description: assessment of the local and systemic adverse reaction within the first 30 days after second vaccination
Time Frame: within the first 30 days after second vaccination
Reporting Status: Not Posted

6. Secondary Outcome: the Safety of Recombinant Hepatitis B Vaccines in Nonresponders
Description: assessment of the local and systemic adverse reaction within the first 30 days after third vaccination
Time Frame: within the first 30 days after third vaccination
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: within 7 months after first dose
Arm/Group | 60mcg/1.0ml Recombinant Hepatitis B Vaccine | 30mcg/1.0ml Recombinant Hepatitis B Vaccine | 10mcg/1.0ml Recombinant Hepatitis B Vaccine
Serious Adverse Events (participants affected / at risk) | 0/434 | 0/435 | 0/222
Other Adverse Events (participants affected / at risk) | 0/434 | 0/435 | 0/222

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No